CLINICAL TRIAL: NCT05017337
Title: A Translational Study of Breast-implant assocIated anaplastIc Large Cell Lymphoma and Capsular Contracture
Brief Title: Breast-implant ASsocIated anaplastIc Large Cell Lymphoma and CApsular Contracture
Acronym: BASILICA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5363; 249930 (Other: IRAS)
Record Dates: First submitted 2021-08-12; First posted 2021-08-23 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Breast Implant-Associated Anaplastic Large Cell Lymphoma; Capsular Contracture, Implant; Breast Implant; Complications
Keywords: BIA-ALCL; Capsular Contracture; Silicone Breast Implants
MeSH Terms: conditions — Implant Capsular Contracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pre- and post-operative blood samples (BASILICA-A prospective, BASILICA-C, BASILICA-N); Capsular tissue samples (BASILICA-C: intra-operative tissue sampling, BASILICA-A retrospective: pathological FFPE blocks); Capsular Washings (BASILICA-C only)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- BASILICA-A: Breast implant associated anaplastic large cell lymphoma (BIA-ALCL) patients recruited both retrospectively and prospectively.
  Pre- and post-operative (3m and 12m) blood samples taken from prospectively recruited patients. Patients undergoing surgery + neo-adjuvant chemotherapy will be invited to donate an additional blood sample following the end of their neo-adjuvant chemotherapy.
  Diagnostic pathology: Where possible fresh seroma aspirate / capsular tissue will be obtained, if not possible the FFPE embedded seroma or tissue block will be requested.
  Post-operative pathological FFPE tissue samples obtained from all recruited patients.
- BASILICA-C: Patients undergoing capsule related surgery (any-grade of capsular contracture, irradiated and unirradiated capsules) recruited prospectively.
  Pre- and post-operative (3m) blood samples taken from all patients. Intra-operative tissue sampling (capsular washings, 2 samples of ADM and 2 samples of non-ADM capsule) from all patients.
- BASILICA-N: Implant naive patients undergoing implant insertion surgery recruited prospectively.
  Pre- and post-operative (3m and 12 m) blood samples taken from all patients.

SUMMARY:
BASILICA is a UK NIHR Biomedical Research Centre funded study recruiting patients at The Royal Marsden NHS Foundation Trust. The study aims to obtain blood and tissue samples from patients with breast implant-associated anaplastic large cell lymphoma (BIA-ALCL), capsular contracture and implant-naïve patients undergoing primary implant insertion surgery for translational scientific analysis.

DETAILED DESCRIPTION:
BASILICA is a translational research study being undertaken at The Royal Marsden NHS Foundation Trust that aims to investigate aetiology of breast implant-associated anaplastic large cell lymphoma (BIA-ALCL), capsular contracture (CC) as well as the immune changes that occur in implant-naïve patients undergoing primary implant insertion surgery.

BIA-ALCL is a rare tumour seen in a very small number of women with textured breast implants. Overall incidence is estimated at 2 per 1,000,000 women/year with a lifetime risk of 1 in 30,000 for textured breast implants. It presents commonly with a sudden seroma around an implant or, occasionally, as a soft tissue mass adjacent to the implant capsule. In 2016, the disease was classified by the WHO as a CD30+ ALK- non-Hodgkin's T-cell lymphoma. Surgery (en bloc capsulectomy) is curative for the majority of cases. Scientific appreciation of aetiology is limited but current thinking implicates chronic inflammation as a protagonist for pathogenesis through hypertonic antigen presentation.

CC is the fibrotic tightening of a capsule that forms around a breast implant and leads to palpable hardening, pain and visible distortion. The biggest risk factor is radiotherapy with quoted incidence rates as high as 50% in some series. Management is a significant clinical challenge with limited options and high recurrence rates. The most common surgical approaches are to remove the capsule (capsulectomy) or exchange and change the anatomical plane of implant placement. The only definitive surgical management is to explant the implant and perform autologous breast reconstruction, if feasible, or, no reconstruction at all.

BASILICA will obtain pathological capsular tissue (CC and BIA-ALCL) and non-pathological capsule tissue (control tissue) as well as blood samples from patients undergoing any form of implant-related surgery. The investigators aim to use these tissues to perform translational analyses investigating the aetiology of each pathology and the physiological immunological response to silicone implant insertion. They hypothesise that 1) specific differences exist in the immunological and matrisomal profiles of CC and BIA-ALCL that drive the pathogenesis of each clinical entity, and that 2) insertion of a silicone prosthesis causes changes in the composition of the humoral and cellular components of the circulating immune system.

ELIGIBILITY:
BASILICA-A

Inclusion Criteria:

1. Patients aged > 16 years
2. Any patient with histopathologically-confirmed ALCL
3. MDT recommendation for capsulectomy
4. Patient consent for capsulectomy

Exclusion Criteria:

1. Inability to give informed consent
2. MDT unable to make recommendation for surgery

BASILICA-C

Inclusion criteria:

1. Patients aged > 16 years
2. Any patient with a capsule arising around an implant, or a clinical diagnosis of capsular contracture
3. MDT recommendation for capsulectomy
4. Patient consent for capsulectomy

Exclusion criteria:

1. Inability to give informed consent
2. MDT unable to make recommendation for surgery#
3. More than one previous implant exchange, or previous extensive capsular surgery

BASILICA-N

Inclusion criteria:

1. Patients aged > 16 years
2. Any patient undergoing implant insertion surgery

Exclusion criteria:

1. Inability to give informed consent
2. MDT unable to make recommendation for surgery
3. Previous implant insertion surgery

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a histopathological diagnosis of BIA-ALCL (BASILICA-A), clinical diagnosis of capsular contracture (BASILICA-C) or implant naive patients undergoing implant insertion surgery (BASILICA-N)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2024-07-27 (Estimated); Study Completion 2024-07-27 (Estimated)

PRIMARY OUTCOMES:
Immunohistochemical analysis of capsular tissue | 3 year following final sample collection
  Perform immunohistochemical profiling of capsular tissues (CC, BIA-ALCL and control) and seroma fluid for immune cell subtypes to determine if differences exist within and between groups (BASILICA A and C).
Capsular tissue profiling using Multi-OMIC technologies | 3 year following final sample collection
  Perform multi-OMIC (methylome, transcriptome, proteome) profiling of capsular tissues (CC, BIA-ALCL and control) to determine if differences exist within and between groups (BASILICA A and C).
Immune profiling of peripheral blood mononuclear cells | 3 year following final sample collection
  Perform immune profiling of peripheral blood mononuclear cells from BIA-ALCL and Non-BIA-ALCL donors (CC and implant naive) to determine if differences exist within and between groups (BASILICA A, C and N)

SECONDARY OUTCOMES:
Appraisal of patient clinical characteristics | 3 year following final sample collection
  Correlate demographic and clinical characteristics of biobank donors with translational scientific dataset (BASILICA A, C and N)

CONTACTS AND LOCATIONS:
Overall Officials: Aadil Khan, FRCS (Plast), Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Royal Marsden Hospital NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No
Non-identifiable patient and translational scientific data may be shared on request with trusted scientific partners.